CLINICAL TRIAL: NCT05396599
Title: A Clinical Study Comparing Postoperative Outcomes Between the TECNIS Intraocular Lens.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision.
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JJSV201EYST
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Eyhance Toric II IOL (Experimental): Model DIU
  Interventions: Device: Model DIU
- TECNIS Synergy Toric II (Experimental): Model DFW
  Interventions: Device: Model DFW
- TECNIS Toric 1-Piece IOL (Active Comparator): Model ZCT
  Interventions: Device: Model ZCT

INTERVENTIONS:
Device: Model DIU — Subjects will be randomized to a treatment group (masked) in ratio 1:1:1. Surgeons will perform standardized, small-incision, cataract surgery and implant the study lenses using a JJSV-validated insertion system qualified for use with the lens to be implanted.
  Arms: Eyhance Toric II IOL
Device: Model DFW — Subjects will be randomized to a treatment group (masked) in ratio 1:1:1. Surgeons will perform standardized, small-incision, cataract surgery and implant the study lenses using a JJSV-validated insertion system qualified for use with the lens to be implanted.
  Arms: TECNIS Synergy Toric II
Device: Model ZCT — Subjects will be randomized to a treatment group (masked) in ratio 1:1:1. Surgeons will perform standardized, small-incision, cataract surgery and implant the study lenses using a JJSV-validated insertion system qualified for use with the lens to be implanted.
  Arms: TECNIS Toric 1-Piece IOL

SUMMARY:
This is a prospective, multi-center, masked, three-arm, randomized clinical study of the TECNIS Eyhance Toric II IOL (test #1) and TECNIS Synergy Toric II (test #2) compared to the TECNIS Toric 1-Piece IOL (control).

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will be enrolled based on surgeon's determination of meeting the minimum study criteria in one or both eyes:

1. Male or female at least 22 years of age
2. Have a cataract in one or both eyes, with planned phacoemulsification and intraocular lens implantation with a toric intraocular lens
3. Regular corneal astigmatism and predicted postoperative residual astigmatism of less than 1.00 D after implantation with a toric intraocular lens in the study eye(s)
4. Availability, willingness and sufficient cognitive awareness to understand the purpose of the examination procedures and comply with postoperative visits
5. Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries.

Exclusion Criteria:

Eligible subjects will be enrolled based on surgeon's determination of meeting the minimum study criteria in one or both eyes:

1. Best-corrected distance visual acuity better than 20/40 Snellen (0.3 logMAR)
2. Potential visual acuity estimated to be worse than 20/32 Snellen (0.2 logMAR)
3. Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery, Including prophylactic peripheral iridotomies and peripheral laser retinal repairs
4. Corneal abnormalities such as stromal, epithelial or endothelial dystrophies (e.g., any observed guttata) that are predicted to cause visual acuity losses to a level worse than 20/30 Snellen during the study
5. Pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils) or unable to dilate to visualize IOL axis (approximately 6.0 mm)
6. Inability to achieve keratometric stability for contact lens wearers (as defined in Section 10.3 Preoperative Procedures)
7. Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
8. Use of systemic or ocular medications that may affect vision
9. Prior, current, or anticipated use during the course of the 6-month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
10. Poorly controlled diabetes
11. Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable.
12. Pregnancy, planned pregnancy, presently lactating, or another condition associated with hormonal fluctuation that could lead to refractive changes
13. Concurrent participation or participation in any other clinical study within 30 days prior to the preoperative visit
14. Any other systemic or ocular disease that, in the opinion of the investigator, may affect the patient's eligibility for the study, affect visual acuity or may require surgical intervention during the study (e.g., macular degeneration, cystoid macular edema, diabetic retinopathy, etc.).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (5):
- United States (5):
  - Shultz Chang Vision, Los Angeles, California
  - Coastal Vision, Orange, California
  - Pacific Eye Associates, A Medical Corporation, San Francisco, California
  - Aloha Vision Consultants, Honolulu, Hawaii
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 subjects were consented. Out of 37 subjects, 2 subjects were screen failures and 35 subjects were enrolled and completed the study.
  Out of 35 subjects, 11 subjects were treated with Test Lens 1 (TECNIS Eyhance Toric II IOL), 13 subjects were treated with Test Lens 2 (TECNIS Synergy Toric II IOL), and 11 subjects were treated with control lens (TECNIS Toric 1-Piece IOL).
Groups:
- Test Lens 1: TECNIS Eyhance Toric II IOL
- Test Lens 2: TECNIS Synergy Toric II IOL
- Control Lens: TECNIS Toric 1-Piece IOL
Period: Overall Study
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens
Started | 11 | 13 | 11
Completed | 11 | 13 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eye
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens | Total
Number analyzed (Participants) | 11 | 13 | 11 | 35
Number analyzed (Eye) | 19 | 22 | 17 | 58
Age, Customized [Number; unit: Years]
  <60 | 2 | 2 | 0 | 4
  60-69 | 2 | 7 | 3 | 12
  70-79 | 5 | 3 | 7 | 15
  >=80 | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 23
  Male | 3 | 5 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 2 | 7 | 10
  Ethnicity: Not Hispanic or Latino | 10 | 11 | 4 | 25
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3 | 8 | 4 | 15
  Caucasian | 7 | 4 | 5 | 16
  Black | 1 | 0 | 0 | 1
  Other | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Rotational Stability of IOL
Description: The percentage of eyes with rotational stability of the IOL at postoperative 1 month.
Time Frame: 1 month
Population: All eyes with available data at 1 month visit.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens
Number analyzed (Participants) | 11 | 13 | 10
Number analyzed (Eyes) | 19 | 22 | 16
Eyes | 19 | 22 | 16

ADVERSE EVENTS:
Time Frame: During the course of the study until termination, 6 months.
Description: All adverse events (AEs), ocular and non-ocular, were monitored/assessed and planned to be reported per subjects.
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT05396599/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT05396599/SAP_001.pdf